CLINICAL TRIAL: NCT06722859
Title: Comparison Between The Results of Open and Microsurgical Decompression in Degenerative Spinal Canal Stenosis in Lumbar Spine in Assuit University Hospital
Brief Title: Comparison Between The Results of Open and Microsurgical Decompression in Degenerative Spinal Canal Stenosis in Lumbar Spine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shamel Mahmoud, Resident of orthopedic and trauma surgery Assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lumbar canal stenosis
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Degenerative Lumbar Canal Stenosis

STUDY DESIGN:
Intervention Model Description: To compare the outcomes of open and microsururgical decompression in degenerative spinal stenosis in lumbar spine
Who Masked: Outcomes Assessor
Masking Description: To compare the outcomes of open and microsururgical decompression in degenerative spinal stenosis in lumbar spine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open surgical decompression (Other)
  Interventions: Procedure: Open surgical decompression in degenerative lumbar canal stenosis; Procedure: Microsurgical decompression
- Microsurgical decompression (Other)
  Interventions: Procedure: Open surgical decompression in degenerative lumbar canal stenosis; Procedure: Microsurgical decompression

INTERVENTIONS:
Procedure: Open surgical decompression in degenerative lumbar canal stenosis — Open surgical decompression in degenerative lumbar canal stenosis
Procedure: Microsurgical decompression — Microsurgical decompression of degenerative lumbar canal stenosis

SUMMARY:
To compare the outcomes of open and microsururgical decompression in degenerative spinal stenosis in lumbar spine

DETAILED DESCRIPTION:
Lumbar spinal stenosis is defined as a circumscribed, osteoligamentous narrowing of the spinal canal. The clinical burden includes backaches and symptoms in the legs that deteriorate upon standing and walking (neurogenic claudication). Lumbar spinal stenosis is the most common cause of lumbar spine diseases in patients > 65 years old requiring surgical treatment; it is estimated that ∼0.1% of the population will need some procedure to treat degenerative lumbar spine conditions. Surgical treatment for lumbar spinal stenosis is indicated in cases of conservative treatment failure. It is also indicated in cases with very acute symptoms and radicular involvement associated with dermatome sensorial and motor changes and progressive worsening of severe neurogenic claudication. Vertebral canal decompression can be performed with several techniques. The gold standard is the open technique with laminectomy or laminotomy, in which laminae are resected or opened; next, the ligamentum flavum, usually thickened, is resected, exposing the nervous structures under compression. Laminotomy can be unilateral, bilateral or divide the spinous process. Damaging the paraspinal muscles and liberal removal of posterior bone may cause iatrogenic spinal instability. The Microsurgical spinal canal decompression decreases paravertebral musculature injury, reducing postoperative complications related to hematomas, seromas and infections and trunk extensor musculature atrophy. The dural sac is decompressed after its exposure and removed to allow the resection of the lateral recess and foramen opening to decompress an adjacent and/or emerging nerve root. It is believed that MIS may limit surgery-related morbidity and mortality by reducing the degree of surgical trauma while maintaining similar surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

patients present with degenerative lumber spinal canal stenosis in one or two level

Exclusion Criteria:

1. degenrative listhesis.
2. degenerative scoliosis.
3. other secondary causes of lumber canal stenosis as tumor , abscesses and infection.
4. Patients with previous lumbar operation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Clincal evaluation by visual analogue scale back pain and leg pain | 12 months